CLINICAL TRIAL: NCT03651687
Title: Guangzhou Surveillance and Clinical Study in Microcephaly
Brief Title: Guangzhou Surveillance and Clinical Study in Microcephaly (GSCSM)
Status: Completed | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Collaborators: Guangzhou Huadu Women and Children Health Care Hospital (Unknown); Guangzhou Liwan Women and Children Health Care Hospital (Unknown); Institut Pasteur (Industry)
Responsible Party: Principal Investigator, Xiu Qiu, Director of the Born in Guangzhou Cohort Study, Guangzhou Women and Children's Medical Center
Other Study IDs: 2016111865-2; 81673181 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2018-08-22; First posted 2018-08-29 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Microcephaly
Keywords: Head circumference; Neurodevelopment; Newborn; Infant; Surveillance; Prediction
MeSH Terms: conditions — Microcephaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At birth: cord, cord blood and placenta; During infancy: oral swab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other:

SUMMARY:
Screening for microcephaly is important at birth and during early childhood. The Guangzhou Surveillance and Clinical Study in Microcephaly (GSCSM) aims to establish a multicentric surveillance system for microcephaly in newborns and infants, to develop a new head circumference reference and microcephaly criteria basing on the local population in Guangzhou, to improve the prediction model of microcephaly, and to follow up the outcomes of the children diagnosed with microcephaly.

DETAILED DESCRIPTION:
Microcephaly is associated with neurological dysfunctions in infants and children. There is not a uniform diagnostic criteria for microcephaly. The World Health Organization (WHO) recommended a criteria of head circumference (HC) less than 2 standard deviations (SD) below the mean of the Intergrowth-21 standard, which was found not applicable to the newborns and infants in Guangzhou.In the GSCSM, the HC measures of newborns are conducted by trained midwives using a standard tool, and extensive information including adverse perinatal outcomes are collected. Longitudinal follow up of infants' neurodevelopment in cognitive, motor, emotional and other domains are also to be conducted. The GSCSM intends to find out the infants who are 'real microcephaly' and most at risk of short-term or long-term adverse outcomes in Guangzhou.

ELIGIBILITY:
Inclusion Criteria:

1. Newborns born after 24+0 weeks of gestation
2. Newborns delivered at the study hospitals

Exclusion Criteria:

1. With major congenital abnormalities
2. Multiple births

Max Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population are infants born in the maternity hospitals from Guangzhou surveillance system.
Sampling Method: Non-Probability Sample
Enrollment: 47369 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Prevalence of microcephaly | At birth
  Assessed by the head circumference measured using a standard tool

SECONDARY OUTCOMES:
Neurodevelopmental performance of children | At birth, 6 weeks, 6 months, 1 year and 2 years
  Including adaptive, gross motor, fine motor, language, and social function; assessed using Gesell Developmental Schedules or Ages and Stages Questionnaire
Head circumference changes of children | At birth, 6 weeks, 6 months, 1 year to 2 years
  Head circumference changes from birth to infancy (catch-up or drop)

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Qiu, MD,PhD, Principal Investigator — Guangzhou Women and Children's Medical Center, China
Locations (1):
- Guangzhou Women and Children's Medical Center, China, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] He JR, Li WD, Lu MS, Guo Y, Chan FF, Lu JH, Zhang LF, Shen SY, Xia XY, Wang P, Mo WJ, Lam KBH, Hirst JE, Xia HM, Qiu X. Birth weight changes in a major city under rapid socioeconomic transition in China. Sci Rep. 2017 Apr 21;7(1):1031. doi: 10.1038/s41598-017-01068-w. PMID 28432291